CLINICAL TRIAL: NCT07041424
Title: Effects of Rebonding Technique and Final Cure on Post-Operative Hypersensitivity in Class 1 Composite Restorations
Brief Title: Effects of Rebonding Technique and Final Cure in Post-operative Hypersensitivity in Class 1 Composite Restorations
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Principal Investigator, Shoaib Rahim, Associate professor, Foundation University Islamabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FUCDOP2501
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Post-Operative Hypersensitivity
Keywords: Rebonding Technique, Post-Operative Hypersensitivity, Composite Restorations

STUDY DESIGN:
Intervention Model Description: four groups. 2 control groups and 2 treatment groups. In group 1, total etch type bonding agent used but no rebonding done. In group 2, total etch bonding agent used and rebonding technique carried out. In group 3, self etch type bonding agent used but no rebonding done. in group 4, self etch bonding agent used and rebonding technique carried out.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group 1: total etch bonding agent without rebonding (Other): composite restoration carried out using total etch bonding agent and no rebonding technique is done
  Interventions: Procedure: treatment group 1: total etch bonding agent used with rebonding technique
- Control group 2: self etch bonding agent without rebonding (Other): composite restoration carried out using self etch bonding agent and no rebonding technique is done
  Interventions: Procedure: treatment group 2: self etch bonding agent used with rebonding technique

INTERVENTIONS:
Procedure: treatment group 1: total etch bonding agent used with rebonding technique — class 1 composite restoration is done using total etch type bonding agent and rebonding technique applied
  Arms: control group 1: total etch bonding agent without rebonding
Procedure: treatment group 2: self etch bonding agent used with rebonding technique — class 1 composite restoration is done using self etch type bonding agent and rebonding technique applied
  Arms: Control group 2: self etch bonding agent without rebonding

SUMMARY:
Rebonding technique has been suggested to address the issue of post-operative hypersensitivity in composite restorations. it involves the application of bonding agent on composite restoration following finishing and polishing.

DETAILED DESCRIPTION:
Rebonding technique has been suggested to address the issue of post-operative hypersensitivity in composite restorations. it involves the application of bonding agent on composite restoration following finishing and polishing. bonding agent fills the gap formed by polymerization shrinkage and hence prevent post-operative hypersensitivity

ELIGIBILITY:
Inclusion Criteria:

* class 1 carious lesion in premolar and molars clinically diagnosed as moderate occlusal caries extending up to middle third of dentin no caries on any other surface of tooth patients with sign and symptom of reversible pulpitis like sharp pain, sensitivity to hot and cold and sweet stimuli lasting foe few seconds

Exclusion Criteria:

* history of generalized sensitivity cavities extending up to pulpal third of dentin cavities need to be restored with direct or indirect pulp capping poor oral hygiene or periodontal disease bruxism and other wear facets chronic anti inflammatory, analgesics or psychotropic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Post-operative hypersensitivity | from treatment to 24 hours and 1 week
  Numeric pain intensity scale 0= no sensitivity 1-3= mild sensitivity 4-6= moderate sensitivity 10=worst possible sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Islamabad, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tekce N, Demirci M, Gokturk SA, Tuncer S, Ozel E, Pala K, Baydemir C. The effect of bonding and surface sealant application on postoperative sensitivity from posterior composites. J Istanb Univ Fac Dent. 2015 Oct 21;49(3):1-10. doi: 10.17096/jiufd.33921. eCollection 2015. PMID 28955539
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28955539/
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/28955539/